CLINICAL TRIAL: NCT04725695
Title: Preoperative Viscous Lidocaine for Upper Gastrointestinal Endoscopy - a Blinded, Randomized, Placebo-controlled Clinical Trial
Brief Title: Preoperative Viscous Lidocaine for Upper Gastrointestinal Endoscopy
Acronym: LIDOGAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of ressources
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Erling Oma, Principal investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020-005177-27
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Anesthetics, Local; Esophagogastroduodenoscopy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viscous lidocaine (Experimental): Oral viscous lidocaine 20 mg/ml, 10 ml
  Interventions: Drug: Viscous Lidocaine
- Placebo (Placebo Comparator): Oral viscous solution without active drug, 10 ml
  Interventions: Drug: Viscous Lidocaine

INTERVENTIONS:
Drug: Viscous Lidocaine — The patients will be randomized to either viscous lidocaine or placebo

SUMMARY:
In this randomized placebo-controlled clinical trial, patients will be randomized to be administered viscous lidocaine or placebo preoperatively to elective upper GI endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to and found fit for upper GI endoscopy in an out patient setting
* Between 18 and 75 years old
* Speaks and understands Danish

Exclusion Criteria:

* Patients admitted for upper GI endoscopy in an in-patient setting
* Patients with dementia and/or other cognitive dysfunction disorders
* Patients primarily complaining of dysphagia
* Patients allergic to lidocaine
* Patients with suspected retention
* Patients who will undergo upper GI endoscopy with nurse-assisted propofol sedation
* Patients who will undergo upper GI endoscopy with assistance of anesthesia-personnel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Ease of intubation | Immediately after the procedure
  The endoscopist will rate the difficulty of intubating the esophagus on a numeric rating scale (NRS) from 0 (worst) to 10 (best)

SECONDARY OUTCOMES:
Ease of examination | Immediately after the procedure
  The endoscopist will rate the difficulty of performing the endoscopy on a numeric rating scale (NRS) from 0 (worst) to 10 (best)
Number of intubation attempts | Peroperatively counted by the assisting nurse
  Total number of intubation attempts until the esophagus is reached
Number of gag reflexes | Peroperatively counted by the assisting nurse
  Total number of gag reflexes during the examination
Patient's perception of discomfort | Immediately after the procedure
  The patient's self-evaluation of discomfort during the examination on a numeric rating scale (NRS) from 0 (worst) to 10 (best)
Patient's willingness to be reexamined | Immediately after the procedure
  The patient's willingness to have the procedure performed again in the future on a numeric rating scale (NRS) from 0 (worst) to 10 (best)
Sedation 1 | Peroperatively
  Number of milligrams midazolam administered during the procedure
Sedation 2 | Peroperatively
  Number of milligrams alfentanil administered during the procedure
Perception of gag reflexes | Immediately after the procedure
  The endoscopist's rating of the patient's degree of gag reflexes, numeric rating scale (NRS) from 0 (worst) to 10 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Erling Oma, MD, PhD, Principal Investigator — Digestive Disease Center, Bispebjerg Hospital
Locations (1):
- Department of Endoscopy, Digestive Disease Center, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After publication for 10 years
Access Criteria: On demand